CLINICAL TRIAL: NCT06726226
Title: Multicenter Cohort for Respiratory Outcome of Preterm Infants
Brief Title: Extremely Preterm Respiratory Outcome Cohort
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); Samsung Medical Center (Other); Seoul National University Bundang Hospital (Other); Chonnam National University Hospital (Other); Severance Hospital, Yonsei University College of Medicine (Unknown); Ajou University Medical Center (Unknown)
Responsible Party: Principal Investigator, Seung Han Shin, Professor, Seoul National University Hospital
Other Study IDs: EPRO
Record Dates: First submitted 2024-01-16; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Infant, Premature; Respiratory Disease
MeSH Terms: conditions — Premature Birth; Respiration Disorders | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples Without DNA — 1. Transtracheal aspirate Collection Timing: Immediately after registration, 3(±1) days after the first collection, 14(±2) days after birth, and 28(±2) days after birth.
  2. Urine Collection Timing: Immediately after registration, 3(±1) days after the first collection, 14(±2) days after birth, and 28(±2) days after birth.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Respiratory cohort: Preterm infants with a gestational age less than 29 weeks
  Interventions: Other: Standard care for preterm infants

INTERVENTIONS:
Other: Standard care for preterm infants — Standard care for preterm infants according to the institutional protocol

SUMMARY:
This study examines the respiratory outcomes of preterm infants born at gestational ages less than 29 weeks, spanning from birth to 24 months corrected age. It delves into the intricacies of respiratory function impairment attributable to diverse factors, such as respiratory distress syndrome, bronchopulmonary dysplasia, postnatal corticosteroids, ventilatory support, as well as nutritional aspect during NICU stay. Furthermore, it scrutinizes the incidence of chronic respiratory diseases stemming from these conditions, assessing their long-term impact on respiratory prognosis post-discharge. In addition to respiratory aspects, the research extends its focus to the growth and developmental outcomes of preterm infants. By synthesizing these multifaceted elements, the study aspires to enhance current treatments and preventative measures for respiratory conditions in preterm infants.

DETAILED DESCRIPTION:
The purpose of this study is to identify various neonatal and perinatal factors that influence the respiratory outcomes of premature infants born at gestational ages less than 29 weeks. Ultimately, the study aims to improve the prevention and treatment of chronic respiratory diseases in these infants by detecting and treating high-risk groups early. Specifically, it seeks to identify factors related to chronic respiratory diseases through the analysis of neonatal specimens.

Despite rising survival rates for premature infants, respiratory complications among these survivors are also increasing. However, there has been no clear identification of factors associated with post-prematurity respiratory diseases. Consequently, there is a growing demand among healthcare professionals in South Korea for respiratory cohorts similar to the PROP cohort in the United States and the Saitama cohort in Japan.

In the Korean Neonatal Network, data is collected on the clinical course during hospitalization and post-discharge growth and development of very low birth weight infants (weighing less than 1500g at birth) admitted to neonatal intensive care units. However, there is currently no information available on respiratory-related diseases, and investigations regarding respiratory outcomes are not being conducted. Therefore, this study aims to analyze the factors associated with respiratory outcomes in preterm survivors and to establish strategies for their prevention and treatment.

According to the research protocol, we are seeking parental consent to enroll preterm infants born before 29 weeks of gestation in participating healthcare institutions within 7 days of their birth. This enrollment will involve collecting biological materials and clinical data to establish a comprehensive database. Clinical data will primarily be obtained by reviewing medical records during the infants' hospitalization period. The assessment of long-term respiratory complications will involve conducting surveys with parents when the infants reach 4, 8, and 12 months of corrected age. Additionally, data collection at 12 and 24 months of corrected age will rely on reviewing medical records from outpatient visits to pediatric and adolescent clinics, based on examination findings and test results. In cases where obtaining in-person follow-up information is challenging, growth and developmental data may be gathered through various means, including telephone calls, text messages, emails, web surveys, and other communication methods. Web survey links will be distributed through text messages.

The primary outcome of this study is to assess the respiratory condition of preterm infants, including evaluating respiratory symptoms, the use of respiratory medications, and hospitalizations related to respiratory diseases. This assessment will be conducted at specific time points: 4, 8, 12, 18, and 24 months of corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at gestational age less than 29 weeks with cohort consent obtained within 7 days of birth

Exclusion Criteria:

* death within 3 days of birth
* severe structural heart defects
* structural abnormalities in the upper airway, lungs, or chest
* congenital anomalies that may impact cardiopulmonary function
* follow-up is difficult until 24 months of age

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study is a multicenter cohort study conducted by a total of 7 institutions (Seoul National University Hospital, Severance Hospital, Asan Medical center, Samsung Medical Hospital, Ajou University Hospital, Bundang Seoul National University Hospital, Chonnam National University Hospital) jointly. It includes all preterm infants born at these hospitals from March 2022 to December 2024, who are born at a gestational age of less than 29 weeks and are admitted to the neonatal intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Postprematurity respiratory disease | 12 months of corrected age
  1. Severe
     * ≥2 respiratory hospitalizations,
     * home supplemental O2 after 3 months or any home mechanical ventilation,
     * systemic steroid exposure or pulmonary vasodilators, or symptoms despite -inhaled corticosteroid use
  2. Mild to moderate
     * one hospitalization
     * home oxygen <3 months corrected age or tracheostomy without ventilation,
     * any inhaled corticosteroid or bronchodilator exposure, or symptoms in ≥2 questionnaires
  3. No/minimal - all other cases
  1. Respiratory medications 2. Hospitalizations for cardiopulmonary cause 3. Coughing, wheezing, or other respiratory symptoms 4. Home technology dependence

SECONDARY OUTCOMES:
Growth assessment | at 24 months of corrected age
  Weight z-score for sex and age based on WHO growth curve
Any delay in developmental scale evaluation | at 24 months of corrected age
  Any delay (<85) in Bayley Scales of Infant and Toddler Development of
  1. Mental Development Index or Psychomotor Development Index in Edition II
  2. Cognitive, Language or Motor domain in Edition III
Long-term respiratory outcome | at 6 years of corrected age
  FEV1 (forced expiratory volume in one second) in pulmonary function test

CONTACTS AND LOCATIONS:
Overall Officials: Seung Han Shin, MD, PhD, Principal Investigator — Seoul National University Children's Hospital
Locations (1):
- Seung Han Shin, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No